CLINICAL TRIAL: NCT03335267
Title: Phase II Trial of CPX (Cytarabine:Daunorubicin) Liposome Injection in Patients >/=60 Years of Age With AML Previously Untreated By Intensive Chemotherapy
Brief Title: Investigator Initiated Trial of CPX-351 for Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510016710
Record Dates: First submitted 2017-09-07; First posted 2017-11-07 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-351 (Cytarabine:Daunorubicin) Injection (Experimental): Dosing for first induction: CPX-351
  • CPX-351 at 100u/m2 will be administered on study days 1, 3 and 5
  Dosing for second induction:
  • CPX-351 at 100 u/m2 will be administered on days 1 and 3
  Dosing for consolidation:
  • CPX-351 at 65 u/m2 will be administered on days 1 and 3
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — Cytarabine:Daunorubicin Liposome Injection

SUMMARY:
This is an open label study to assess the suitability of CPX-351 as first intensive therapy in elderly (age ≥60 years) patients with AML. Patients may have received prior AML treatment with non-intensive regimens, e.g. hypomethylating agents, low dose Ara C or lenolidomide, but may not have received intensive AML treatment with anthracyclines and/or cytarabine prior to enrollment on this trial. The outcome of elderly patients following intensive treatment with CPX-351 will be measured by clinical endpoints for efficacy and safety and by biological/functional response.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily give informed consent
* Age≥60 years at the time of study treatment
* Pathological diagnosis of AML according to WHO criteria (with >20% blasts in the peripheral blood or bone marrow) including:
* De novo AML with normal karyotype or adverse karyotypes (including patients with karyotypic abnormalities characteristic of MDS)
* Secondary AML: transformed from prior MDS or MPN, confirmed by bone marrow documentation of prior antecedent hematologic disorder
* Therapy-related AML: t-AML, requires documented history of prior cytotoxic therapy or ionizing radiotherapy for an unrelated disease
* Performance status >50% KPS, ECOG 0-2
* Laboratory values fulfilling the following:
* Serum creatinine < 2.5 mg/dL
* Serum total bilirubin < 2.5 mg/dL,
* Serum alanine aminotransferase or aspartate aminotransferase < 3 times the ULN
* Patients with elevated liver enzymes and serum creatinine values secondary to AML are eligible after discussion with PI
* Cardiac ejection fraction ≥ 50% by echocardiography or MUGA
* Patients with history of second malignancies in remission may be eligible if there is clinical evidence of disease stability off cytotoxic chemotherapy, documented by imaging, tumor marker studies, etc., at screening. Patients maintained on long-term non-chemotherapy treatment, e.g., hormonal therapy, are eligible.

Exclusion Criteria:

* Acute promyelocytic leukemia [t(15;17)]
* Clinical evidence of active CNS leukemia
* Prior intensive chemotherapy for AML with anthracycline/cytarabine-based regimens and/ or prior HSCT. Patients may have been treated with commercially available or investigational hypomethylating agents (e.g. decitabine, azacitidine, SGI-110), lenalidomide, or low-dose cytarabine (not to exceed 20 mg/m2 daily for 14 days for ≤ 6 cycles)
* Prior treatment including HMA, systemic chemotherapy, surgery, or radiation therapy must have been completed at least 7 days before start of study treatment or after discussion with PI. Treatment with investigational agents must have been completed at least 14 days prior to study drug treatment. Hydroxyurea is permitted for control of blood counts before the start of study treatment. Toxicities associated with prior therapies must have recovered to grade 1 or less prior to start of study treatment.
* Patients with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent).
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent
* Patients with myocardial impairment of any cause (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging)
* Active or uncontrolled infection. Patients with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥72 hrs.
* Patients with current or recent evidence of invasive fungal infection (blood or tissue culture); patients with recent fungal infection must have a subsequent negative cultures to be eligible
* Known HIV (new testing not required) or evidence of active hepatitis B or C infection (with rising transaminase values)
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-metabolism disorder
* History of prior bone marrow or solid organ transplantation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen K Ritchie, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CPX-351 (Cytarabine:Daunorubicin) Injection: Dosing for first induction: CPX-351
  • CPX-351 at 100u/m2 will be administered on study days 1, 3 and 5
  Dosing for second induction:
  • CPX-351 at 100 u/m2 will be administered on days 1 and 3
  Dosing for consolidation:
  • CPX-351 at 65 u/m2 will be administered on days 1 and 3
  CPX-351: Cytarabine:Daunorubicin Liposome Injection
Period: Overall Study
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: Years] | 70.98 [60 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: Participants]
  United States | 30
Newly Diagnosed AML Patients Aged ≥ 60 Years [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy
Description: Overall survival is measured from the date of registration to death from any cause. Patients not known to have died will be censored on the date they were last known to be alive. Patients were followed for 2.5 years.
Time Frame: 2.5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
Number analyzed (Participants) | 30
Participants | 7

2. Primary Outcome: 30-Day Mortality Rate
Description: Mortality rate at Day 30
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
Number analyzed (Participants) | 30
Participants | 2

3. Secondary Outcome: Complete Response Rate (CR, CRp, CRi, and CR+CRp+CRi)
Description: The number of patients who achieve response will be divided by the number of patients in the efficacy population to determine response rate.
Time Frame: 30 days post-treatment, up to 3 months post-baseline
Population: 14 subjects were excluded from analysis for this measure due to treatment failure (progressive disease or non-evaluable).
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
Number analyzed (Participants) | 16
Participants
  Complete remission (CR) | 11
  Complete remission with incomplete recovery (CRi) | 5

4. Secondary Outcome: Change in Relationship of Cognitive Function to Treatment Response and OS, Event-free Survival and Morphologic Leukemia Free State as Measured by the MOCA
Description: The Montreal Cognitive Assessment (MOCA) is a 30-point test which assesses several cognitive domains. Possible total scores range from 0 to 30. The results can be interpreted as follows: normal cognition: 26-30 points, mild cognitive impairment: 18-25 points, moderate cognitive impairment: 10-17 points, and severe cognitive impairment: under 10 points.
Time Frame: Screening through 30 days post-treatment, up to 3 months post-baseline
Population: 9 subjects did not complete the MOCA and they were excluded from analysis for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
Number analyzed (Participants) | 21
score on a scale
  Montreal Cognitive Assessment (baseline) | 24.72 (2.85)
  Montreal Cognitive Assessment (30 days post-treatment) | 25.79 (2.99)

5. Secondary Outcome: Change in Relationship of Cognitive Function to Treatment Response and OS, Event-free Survival and Morphologic Leukemia Free State as Measured by the Blessed Orientation-Memory-Concentration Test
Description: The Blessed Orientation-Memory-Concentration Test is designed to evaluate older patients for early dementia. Possible total scores range from 0 (all items answered correctly) to 28 (all items answered incorrectly).
Time Frame: Screening through 30 days post-treatment, up to 3 months post-baseline
Population: 9 subjects did not complete the Blessed Orientation-Memory-Concentration Test and they were excluded from analysis for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
Number analyzed (Participants) | 21
score on a scale
  Blessed Orientation-Memory-Concentration Test (baseline) | 3.45 (2.87)
  Blessed Orientation-Memory-Concentration Test (30 days post-treatment) | 2 (2.27)

6. Secondary Outcome: Incidence of Adverse Events
Description: Adverse events included neutropenic fever, transient episodes of pericarditis, febrile neutropenia, streptococcus bacteremia, hypotensive episode, severe diffuse cerebral dysfunction, UTI (klebsiella pneumonia), anorexia with malnutrition, hypophosphatemia, hypokalemia, purple macules, elevated ALT, hypoalbuminemia, hyperbilirubinemia, syncope, joint pain, transaminitis, bacteremia, typhlitis, VRE bacteremia, Osteomyelitis, Decreased LVEF, GI adenovirus, Acute kidney injury, pulmonary edema, neutropenia, bronchospasm, bone pain, urinary incontinence, c. difficile infection, mucositis, and vaginal pain.
Time Frame: Through treatment completion, an average of 1 year
Measure: Number; unit: events
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
Number analyzed (Participants) | 30
events | 56

ADVERSE EVENTS:
Time Frame: 2.5 Years
Arm/Group | CPX-351 (Cytarabine:Daunorubicin) Injection
All-Cause Mortality (participants affected / at risk) | 23/30
Serious Adverse Events (participants affected / at risk) | 14/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-351 (Cytarabine:Daunorubicin) Injection (N=30)
Neutropenic fever (General disorders) | 2
Hemorrhagic cerebrovascular accident (Vascular disorders) | 1
Septic shock (Infections and infestations) | 1
Volume overload (Cardiac disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 2
Massive hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Ejection fraction decreased (Cardiac disorders) | 6
Failure to thrive (General disorders) | 1
Cardiopulmonary arrest (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-351 (Cytarabine:Daunorubicin) Injection (N=30)
Neutropenic fever (General disorders) | 7
Transient episodes of pericarditis (Cardiac disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 12
Streptococcus bacteremia (Infections and infestations) | 1
Hypotensive episode (Vascular disorders) | 1
Severe diffuse cerebral dysfunction (Nervous system disorders) | 1
UTI (klebsiella pneumonia) (Infections and infestations) | 1
Anorexia with malnutrition (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Investigations) | 2
Hypokalemia (Investigations) | 3
Purple macules (Skin and subcutaneous tissue disorders) | 1
Elevated ALT (Investigations) | 1
Hypoalbuminemia (Investigations) | 1
Hyperbilirubinemia (Investigations) | 3
Syncope (Nervous system disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Transaminitis (Investigations) | 1
Bacteremia (Infections and infestations) | 1
Typhlitis (Infections and infestations) | 1
VRE bacteremia (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Decreased LVEF (Cardiac disorders) | 2
GI adenovirus (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
C. difficile infection (Infections and infestations) | 1
Mucositis (Gastrointestinal disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
We intended to collect and compare baseline and end of induction data to assess the relationship of cognitive function to treatment response and overall survival, event-free survival, and morphologic leukemia free state. Subjects on treatment were usually too unwell to complete the questionnaires, which resulted in significant missing data. We were unable to determine if the relationship was statistically significant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT03335267/Prot_SAP_000.pdf